CLINICAL TRIAL: NCT04751110
Title: Ultrasound Guided Rhomboid Intercostal Block for Myofascial Pain Syndrome: Observational Study
Brief Title: Ultrasound Guided Rhomboid Intercostal Block for Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Selin Guven Kose, Principal Investigator, Diskapi Teaching and Research Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 98/05
Record Dates: First submitted 2021-02-05; First posted 2021-02-11 (Actual); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Myofascial Pain Syndrome
Keywords: rhomboid intercostal block; ultrasound guided block
MeSH Terms: conditions — Myofascial Pain Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- block group (Other): ultrasound guided rhomboid intercostal block will performed
  Interventions: Other: ultrasound guided rhomboid intercostal block

INTERVENTIONS:
Other: ultrasound guided rhomboid intercostal block — A linear ultrasound probe was medially placed in the sagittal plane on the medial border of the scapula at the T5-T7 level. We inserted a 22-gauge needle into the fascial plane between the rhomboid major and intercostal muscles in a craniocaudal direction and injected 15 ml mixture of 0.25% bupivacaine with 8 mg of dexamethasone into the fascial plane.

SUMMARY:
Rhomboid intercostal block (RIB) is an interfacial plane block described in 2016. It creates analgesia at T2-T9 levels in the hemithorax by applying local anesthetic to the fascia between the rhomboid muscle and the intercostal muscle. It has been used effectively in patients with chronic pain. Recently published report has shown that rhomboid intercostal block (RIB) may provide effective pain control for myofascial pain syndrome (MPS), too. MPS is a regional pain syndrome characterized by trigger points detected in one or more regional muscle groups. The investigators planned a prospective observational study, a total of 30 patients who will apply to our clinic with MPS, will register in research. The investigators will perform ultrasound-guided RIB, and evaluate the clinical outcomes.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MPS) is the most common cause of musculoskeletal pain and its prevalence in the population is reported to be 21-30%. Rhomboid intercostal block (RIB) is an interfacial plane block described in 2016. It creates analgesia at T2-T9 levels in the hemithorax by applying local anesthetic to the fascia between the rhomboid muscle and the intercostal muscle. It has been used effectively in patients with chronic pain. The investigators planned a prospective observational study.From february to march 10 2021, a total of 30 patients who will apply to our clinic with MPS, will register in research. The investigators will perform ultrasound-guided RIB, and evaluate the clinical outcome Ultrasound guided RIB will applied with linear probe, in plane technique. Block needle was inserted to plane between the rhomboid muscle and intercostal muscles over the T5-6 ribs 2 cm to 3 cm medially from the medial border of the scapula. 13ml of bupivacaine 0.25% and 8mg dexamethasone mixture will inject into the fascial plane. Numerical Rating Scale (NRS) will recorded before and after the block at 30 minutes, day 1, 1-2-4-6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Complaint of myofascial pain
* Pain that is rated at least 3 on a numerical rating scale (NRS, 0 = no pain, 10 = the worst pain)

Exclusion Criteria:

* pregnancy
* the presence of coagulopathy, or the use of anticoagulants
* a history of surgery on the block area
* allergic to bupivacaine
* decline to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) Pain Score Change | Change from baseline to minutes 30, day 1, week 1, 2, 4, 6 after the block
  The 11-point NRS consists of numbers between 0 and 10 where 0 indicates "no pain" and 10 indicates "maximum pain." The patient is instructed to identify one number between 0 and 10, which is best representative of their pain intensity.

CONTACTS AND LOCATIONS:
Overall Officials: Selin Guven Kose, Principal Investigator — Diskapi Yildirim Beyazit Education and Research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Training and Research Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Borg-Stein J, Iaccarino MA. Myofascial pain syndrome treatments. Phys Med Rehabil Clin N Am. 2014 May;25(2):357-74. doi: 10.1016/j.pmr.2014.01.012. Epub 2014 Mar 17. PMID 24787338
- [Background] Ekinci M, Ciftci B, Alici HA, Ahiskalioglu A. Ultrasound-guided rhomboid intercostal block effectively manages myofascial pain. Korean J Anesthesiol. 2020 Dec;73(6):564-565. doi: 10.4097/kja.20211. Epub 2020 May 12. No abstract available. PMID 32392670
- [Background] Piraccini E, De Lorenzo E, Maitan S. Rhomboid intercostal block for myofascial pain syndrome in a patient with amyotrophic lateral sclerosis. Minerva Anestesiol. 2019 Dec;85(12):1367-1369. doi: 10.23736/S0375-9393.19.13791-1. Epub 2019 Jul 22. No abstract available. PMID 31334619
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611